CLINICAL TRIAL: NCT06318104
Title: Efficacy and Safety of a Triple Eradication Scheme for Helicobacter Pylori Based on Amoxicillin 1g + Clarithromycin 500 mg and Tegoprazan 50 mg vs Amoxicillin 1g + Clarithromycin 500 mg and Esomeprazole 40 mg Twice a Day for 14 Days
Brief Title: Efficacy and Safety of a Triple Eradication Scheme for Helicobacter Pylori Based on Tegoprazan vs Esomeprazole
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital General de México Dr. Eduardo Liceaga (Other Government)
Responsible Party: Principal Investigator, Yoali Maribel Velasco Santiago, Doctor assigned to gastroenterology, Hospital General de México Dr. Eduardo Liceaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DI/24/310/03/4
Record Dates: First submitted 2024-02-28; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Helicobacter Pylori Infection
Keywords: Tegoprazan; Esomeprazole; Effectiveness; Safety
MeSH Terms: interventions — tegoprazan; Esomeprazole

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tegoprazan Group (Active Comparator): Tegoprazan 50 mg BID for 14 days, amoxicillin 1gr BID for 14 days, clarithromycin 500 mg BID for 14 days
  Interventions: Drug: Tegoprazan
- Esomeprazole Group (Active Comparator): Esomeprazole 40 mg BID for 14 days, amoxicillin 1gr BID for 14 days, clarithromycin 500 mg BID for 14 days
  Interventions: Drug: Esomeprazole 40mg

INTERVENTIONS:
Drug: Tegoprazan — Tegoprazan 50 mg BID + amoxicillin 1 gr BID + clarithromycin 500 mg BID all for 14 days.
  Other Names: P-CAB
  Arms: Tegoprazan Group
Drug: Esomeprazole 40mg — Esomeprazole 40 mg BID + amoxicillin 1 gr BID + clarithromycin 500 mg BID all for 14 days.
  Other Names: PPI
  Arms: Esomeprazole Group

SUMMARY:
In Mexico, quadruple therapy is used to treat Helicobacter pylori (H.P.) at the expense of greater adverse effects, costs, and lower adherence to treatment. According to evidence, a competitive potassium channel blocker (P-CAB) is non-inferior to a proton pump inhibitor (PPI) and can improve the eradication rate of H.P. while maintaining triple therapy antibiotics (amoxicillin-clarithromycin) without increasing adverse effects, fewer drugs and better adherence to treatment. It is proposed to study the effect of a P-CAB in the eradication of H.P. as part of a triple therapy in Mexican patients, assuming that the efficacy and safety of a triple therapy of amoxicillin-clarithromycin-tegoprazan will be superior to amoxicillin-clarithromycin-esomeprazole.

DETAILED DESCRIPTION:
160 patients with a diagnosis of H.P. infection with indication for treatment in accordance with the IV Mexican Consensus on Helicobacter Pylori, evaluated in the Gastroenterology outpatient clinic, will be recruited. Participants will be randomized into two groups, one group will receive tegoprazan 50 mg BID, clarithromycin 500 mg BID and amoxicillin 1 gr BID for 14 days and the second group will receive esomeprazole 40 mg BID, clarithromycin 500 mg BID and amoxicillin 1 gr BID for 14 days. Through complementary studies, telephone calls and application of questionnaires, adherence to treatment will be evaluated and adverse events will be monitored, and once the treatment period is completed, a breath test will be performed between days 28-42 to verify eradication, thereby evaluating effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* First-degree relatives with a history of gastric cancer.
* Clinical diagnosis of uninvestigated dyspepsia in patients under 50 years of age.
* Diagnosis of Gastric Mucosa - Aassociated Lymphoid Tissue (MALT) Lymphoma.
* Iron deficiency anemia.
* Unexplained thrombocytopenic purpura.

Exclusion Criteria:

* Patients who have social coverage.
* Previous eradication treatment for Helicobacter Pylori.
* Acute upper gastrointestinal bleeding and active gastric and/or duodenal ulcer.
* History of surgery that affects gastric acid secretion (vagotomy, gastrointestinal resection).
* Disorders of gastric acid hypersecretion (Zollinger-Ellison Syndrome).
* Any serious hematological, cardiovascular, neurological, nephro-urological, hepatic and pulmonary disorders.
* Pregnancy or lactation.
* Allergy to any of the study medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-04-19 (Estimated); Primary Completion 2024-11-29 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Response to treatment by determining the eradication rate | Two months
  The eradication rate will be measured by a carbon-13 urea breath test that will verify the eradication of Helicobacter pylori. The eradication rate of the triple regimen based on clarithromycin - amoxicillin - esomeprazole vs clarithromycin - amoxicillin - tegoprazan will be compared.
Compared Treatment-related adverse events | Two months
  Treatment-related adverse events will be evaluated by complementary serum studies and interrogated according to system organ classes and preferred terms using MedDRA. Adverse events related to the treatment of the triple regimen based on clarithromycin - amoxicillin - esomeprazole vs clarithromycin - amoxicillin - tegoprazan will be compared.

SECONDARY OUTCOMES:
Brief Medication Questionnaire | Two weeks
  Identify the factors associated with medication consumption, by applying the Brief Medication Questionnaire on day 7 and 14 of treatment, via telephone call and in person.
Percentage of patients with adherence to treatment | Two weeks
  Adherence to treatment will be evaluated by calculating the percentage of compliance and tablet count, which is based on the count of the number of tablets left in the container compared to the amount initially indicated, and the time between the indication and the count. The percentage of adherence to eradication treatment will be compared in patients treated with the scheme based on tegoprazan vs. proton pump inhibitor.
Report all Treatment-related adverse events | Two months
  Treatment-related adverse events will be evaluated by complementary serum studies and interrogated according to system organ classes and preferred terms using MedDRA.

CONTACTS AND LOCATIONS:
Overall Officials: Yoali M Velasco Santiago, Principal Investigator — Hospital General de México Dr. Eduardo Liceaga

IPD SHARING:
Plan to Share IPD: No
For legal confidentiality reasons.

REFERENCES:
- [Background] Leja M, Grinberga-Derica I, Bilgilier C, Steininger C. Review: Epidemiology of Helicobacter pylori infection. Helicobacter. 2019 Sep;24 Suppl 1:e12635. doi: 10.1111/hel.12635. PMID 31486242
- [Background] Torres J, Ferreira RM, Kato I. Editorial: The role of Helicobacter pylori in gastric carcinogenesis. Front Oncol. 2023 Jun 26;13:1233890. doi: 10.3389/fonc.2023.1233890. eCollection 2023. No abstract available. PMID 37434981
- [Background] Porras C, Nodora J, Sexton R, Ferreccio C, Jimenez S, Dominguez RL, Cook P, Anderson G, Morgan DR, Baker LH, Greenberg ER, Herrero R. Epidemiology of Helicobacter pylori infection in six Latin American countries (SWOG Trial S0701). Cancer Causes Control. 2013 Feb;24(2):209-15. doi: 10.1007/s10552-012-0117-5. Epub 2012 Dec 12. PMID 23263777
- [Background] Bosques-Padilla FJ, Remes-Troche JM, Gonzalez-Huezo MS, Perez-Perez G, Torres-Lopez J, Abdo-Francis JM, Bielsa-Fernandez MV, Camargo MC, Esquivel-Ayanegui F, Garza-Gonzalez E, Hernandez-Guerrero AI, Herrera-Goepfert R, Huerta-Iga FM, Leal-Herrera Y, Lopez-Colombo A, Ortiz-Olvera NX, Riquelme-Perez A, Sampieri CL, Uscanga-Dominguez LF, Velarde-Ruiz Velasco JA. The fourth Mexican consensus on Helicobacter pylori. Rev Gastroenterol Mex (Engl Ed). 2018 Jul-Sep;83(3):325-341. doi: 10.1016/j.rgmx.2018.05.003. Epub 2018 Jun 22. English, Spanish. PMID 29941237
- [Background] Li Q. Bacterial infection and microbiota in carcinogenesis and tumor development. Front Cell Infect Microbiol. 2023 Nov 15;13:1294082. doi: 10.3389/fcimb.2023.1294082. eCollection 2023. PMID 38035341
- [Background] Luo S, Ru J, Khan Mirzaei M, Xue J, Peng X, Ralser A, Hadi JL, Mejias-Luque R, Gerhard M, Deng L. Helicobacter pylori infection alters gut virome by expanding temperate phages linked to increased risk of colorectal cancer. Gut. 2024 Aug 8;73(9):1592-1595. doi: 10.1136/gutjnl-2023-330362. No abstract available. PMID 37918887
- [Background] Sun Q, Yuan C, Zhou S, Lu J, Zeng M, Cai X, Song H. Helicobacter pylori infection: a dynamic process from diagnosis to treatment. Front Cell Infect Microbiol. 2023 Oct 19;13:1257817. doi: 10.3389/fcimb.2023.1257817. eCollection 2023. PMID 37928189
- [Background] Shakir SM, Shakir FA, Couturier MR. Updates to the Diagnosis and Clinical Management of Helicobacter pylori Infections. Clin Chem. 2023 Aug 2;69(8):869-880. doi: 10.1093/clinchem/hvad081. PMID 37473423
- [Background] Shah SC, Iyer PG, Moss SF. AGA Clinical Practice Update on the Management of Refractory Helicobacter pylori Infection: Expert Review. Gastroenterology. 2021 Apr;160(5):1831-1841. doi: 10.1053/j.gastro.2020.11.059. Epub 2021 Jan 29. PMID 33524402
- [Background] Chey WD, Leontiadis GI, Howden CW, Moss SF. ACG Clinical Guideline: Treatment of Helicobacter pylori Infection. Am J Gastroenterol. 2017 Feb;112(2):212-239. doi: 10.1038/ajg.2016.563. Epub 2017 Jan 10. PMID 28071659
- [Background] World gastroenterology organisation global guideline: Helicobacter pylori in developing countries. J Dig Dis. 2011 Oct;12(5):319-26. doi: 10.1111/j.1751-2980.2011.00529.x. No abstract available. PMID 21955424
- [Background] Malfertheiner P, Megraud F, Rokkas T, Gisbert JP, Liou JM, Schulz C, Gasbarrini A, Hunt RH, Leja M, O'Morain C, Rugge M, Suerbaum S, Tilg H, Sugano K, El-Omar EM; European Helicobacter and Microbiota Study group. Management of Helicobacter pylori infection: the Maastricht VI/Florence consensus report. Gut. 2022 Aug 8:gutjnl-2022-327745. doi: 10.1136/gutjnl-2022-327745. Online ahead of print. PMID 35944925
- [Background] Malfertheiner P, Camargo MC, El-Omar E, Liou JM, Peek R, Schulz C, Smith SI, Suerbaum S. Helicobacter pylori infection. Nat Rev Dis Primers. 2023 Apr 20;9(1):19. doi: 10.1038/s41572-023-00431-8. PMID 37081005
- [Background] Sugimoto M, Furuta T. Efficacy of tailored Helicobacter pylori eradication therapy based on antibiotic susceptibility and CYP2C19 genotype. World J Gastroenterol. 2014 Jun 7;20(21):6400-11. doi: 10.3748/wjg.v20.i21.6400. PMID 24914361
- [Background] Zhou BG, Yan XL, Wan LY, Zhang Q, Li B, Ai YW. Effect of enhanced patient instructions on Helicobacter pylori eradication: A systematic review and meta-analysis of randomized controlled trials. Helicobacter. 2022 Apr;27(2):e12869. doi: 10.1111/hel.12869. Epub 2022 Feb 18. PMID 35178810
- [Background] Savoldi A, Carrara E, Graham DY, Conti M, Tacconelli E. Prevalence of Antibiotic Resistance in Helicobacter pylori: A Systematic Review and Meta-analysis in World Health Organization Regions. Gastroenterology. 2018 Nov;155(5):1372-1382.e17. doi: 10.1053/j.gastro.2018.07.007. Epub 2018 Jul 7. PMID 29990487
- [Background] Torres J, Camorlinga-Ponce M, Perez-Perez G, Madrazo-De la Garza A, Dehesa M, Gonzalez-Valencia G, Munoz O. Increasing multidrug resistance in Helicobacter pylori strains isolated from children and adults in Mexico. J Clin Microbiol. 2001 Jul;39(7):2677-80. doi: 10.1128/JCM.39.7.2677-2680.2001. PMID 11427594
- [Background] Alarcon-Millan J, Fernandez-Tilapa G, Cortes-Malagon EM, Castanon-Sanchez CA, De Sampedro-Reyes J, Cruz-Del Carmen I, Betancourt-Linares R, Roman-Roman A. Clarithromycin resistance and prevalence of Helicobacter pylori virulent genotypes in patients from Southern Mexico with chronic gastritis. Infect Genet Evol. 2016 Oct;44:190-198. doi: 10.1016/j.meegid.2016.06.044. Epub 2016 Jun 26. PMID 27355861
- [Background] Ng HY, Leung WK, Cheung KS. Antibiotic Resistance, Susceptibility Testing and Stewardship in Helicobacter pylori Infection. Int J Mol Sci. 2023 Jul 20;24(14):11708. doi: 10.3390/ijms241411708. PMID 37511471
- [Background] Mladenova I. Epidemiology of Helicobacter pylori Resistance to Antibiotics (A Narrative Review). Antibiotics (Basel). 2023 Jul 13;12(7):1184. doi: 10.3390/antibiotics12071184. PMID 37508280
- [Background] Gatta L, Vakil N, Vaira D, Scarpignato C. Global eradication rates for Helicobacter pylori infection: systematic review and meta-analysis of sequential therapy. BMJ. 2013 Aug 7;347:f4587. doi: 10.1136/bmj.f4587. PMID 23926315
- [Background] Lima JJ, Thomas CD, Barbarino J, Desta Z, Van Driest SL, El Rouby N, Johnson JA, Cavallari LH, Shakhnovich V, Thacker DL, Scott SA, Schwab M, Uppugunduri CRS, Formea CM, Franciosi JP, Sangkuhl K, Gaedigk A, Klein TE, Gammal RS, Furuta T. Clinical Pharmacogenetics Implementation Consortium (CPIC) Guideline for CYP2C19 and Proton Pump Inhibitor Dosing. Clin Pharmacol Ther. 2021 Jun;109(6):1417-1423. doi: 10.1002/cpt.2015. Epub 2020 Sep 20. PMID 32770672
- [Background] Domingues G, Chinzon D, Moraes-Filho JPP, Senra JT, Perrotti M, Zaterka S. Potassium-competitive acid blockers, a new therapeutic class, and their role in acid-related diseases: a narrative review. Prz Gastroenterol. 2023;18(1):47-55. doi: 10.5114/pg.2022.116673. Epub 2022 Aug 15. PMID 37007753
- [Background] Shah A, Usman O, Zahra T, Chaudhari SS, Mulaka GSR, Masood R, Batool S, Saleem F. Efficacy and Safety of Potassium-Competitive Acid Blockers Versus Proton Pump Inhibitors as Helicobacter pylori Eradication Therapy: A Meta-Analysis of Randomized Clinical Trials. Cureus. 2023 Nov 7;15(11):e48465. doi: 10.7759/cureus.48465. eCollection 2023 Nov. PMID 38074044
- [Background] Echizen H. The First-in-Class Potassium-Competitive Acid Blocker, Vonoprazan Fumarate: Pharmacokinetic and Pharmacodynamic Considerations. Clin Pharmacokinet. 2016 Apr;55(4):409-18. doi: 10.1007/s40262-015-0326-7. PMID 26369775
- [Background] Okamura T, Suga T, Nagaya T, Arakura N, Matsumoto T, Nakayama Y, Tanaka E. Antimicrobial resistance and characteristics of eradication therapy of Helicobacter pylori in Japan: a multi-generational comparison. Helicobacter. 2014 Jun;19(3):214-20. doi: 10.1111/hel.12124. Epub 2014 Apr 3. PMID 24758533
- [Background] Kato M, Ota H, Okuda M, Kikuchi S, Satoh K, Shimoyama T, Suzuki H, Handa O, Furuta T, Mabe K, Murakami K, Sugiyama T, Uemura N, Takahashi S. Guidelines for the management of Helicobacter pylori infection in Japan: 2016 Revised Edition. Helicobacter. 2019 Aug;24(4):e12597. doi: 10.1111/hel.12597. Epub 2019 May 20. PMID 31111585
- [Background] Murakami K, Sakurai Y, Shiino M, Funao N, Nishimura A, Asaka M. Vonoprazan, a novel potassium-competitive acid blocker, as a component of first-line and second-line triple therapy for Helicobacter pylori eradication: a phase III, randomised, double-blind study. Gut. 2016 Sep;65(9):1439-46. doi: 10.1136/gutjnl-2015-311304. Epub 2016 Mar 2. PMID 26935876
- [Background] Choi YJ, Lee YC, Kim JM, Kim JI, Moon JS, Lim YJ, Baik GH, Son BK, Lee HL, Kim KO, Kim N, Ko KH, Jung HK, Shim KN, Chun HJ, Kim BW, Lee H, Kim JH, Chung H, Kim SG, Jang JY. Triple Therapy-Based on Tegoprazan, a New Potassium-Competitive Acid Blocker, for First-Line Treatment of Helicobacter pylori Infection: A Randomized, Double-Blind, Phase III, Clinical Trial. Gut Liver. 2022 Jul 15;16(4):535-546. doi: 10.5009/gnl220055. Epub 2022 Jul 6. PMID 35791797
- [Background] Sakurai Y, Nishimura A, Kennedy G, Hibberd M, Jenkins R, Okamoto H, Yoneyama T, Jenkins H, Ashida K, Irie S, Taubel J. Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Rising TAK-438 (Vonoprazan) Doses in Healthy Male Japanese/non-Japanese Subjects. Clin Transl Gastroenterol. 2015 Jun 25;6(6):e94. doi: 10.1038/ctg.2015.18. PMID 26111126
- See also: Review: Global Cancer Observatory — https://gco.iarc.fr/